CLINICAL TRIAL: NCT06298266
Title: Clinical Study to Evaluate the Safety, Tolerability and Initial Efficacy of Anti-GPRC5D-CD19-CAR-T in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: To Assess Safety, Tolerability, and Efficacy of Anti-GPRC5D-CD19-CAR-T in Relapsed/Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangdong Second Provincial General Hospital (Other)
Responsible Party: Principal Investigator, Qing Zhang, Chief Physician, Guangdong Second Provincial General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GD2H-XYK-001
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: GPRC5D-CD19 CART; Multiple myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- infusion of GPRC5D-CD19 CAR T injection (Experimental): Infusion of GPRC5D-CD19 CAR T cells injection by dose of 1.0×10^6 /kg±20 % CAR-T ，3.0×10^6 /kg±20%、6.0×10^6 /kg±20%. Administration method: intravenous infusion. Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion.
  Interventions: Biological: infusion of GPRC5D-CD19 CAR T injection

INTERVENTIONS:
Biological: infusion of GPRC5D-CD19 CAR T injection — Infusion of GPRC5D-CD19 CAR T cells injection by dose of 1.0×10^6 /kg±20 % CAR-T ，3.0×10^6 /kg±20%、6.0×10^6 /kg±20%. Administration method: intravenous infusion. Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
To evaluate the safety and tolerability of anti-GPRC5D-CD19 CAR-T cells infusion in subjects with relapsed and refractory multiple myeloma

DETAILED DESCRIPTION:
This study is a single-arm, single-center clinical study of IIT to evaluate the safety, tolerability, pharmacokinetic profile, and initial efficacy of GPRC5D-CD19 CAR T cells in subjects with MM. The safety of GPRC5D-CD19 CAR T was evaluated by observing adverse events after cell therapy. Evaluate the effectiveness of GPRC5D-CD19 CAR T treatment compared to the results of the subjects' own previous standard treatment regimens or base data. Blood and bone marrow were collected before and 24 months after the GPRC5D-CD19 CAR T infusion to detection.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient or their legal guardian understands and voluntarily signs the informed consent form and is expected to complete the follow-up examinations and treatments.

  2. Age between 18-75 years, regardless of gender. 3. Diagnosed with multiple myeloma according to the IMWG diagnostic criteria, and GPRC5D expression in bone marrow is positive (>10%).

  4. Has failed treatment with at least three different mechanisms of drugs (including chemotherapy, proteasome inhibitors, immune modulators, etc.), or has experienced disease progression or relapse within 6 months after the last treatment.

  5. Measurable lesions are present based on any of the following criteria during screening: (1) Serum monoclonal immunoglobulin (M-protein) level ≥1.0 g/dL; (2) Urine M-protein level ≥200 mg/24 hours; (3) Diagnosed with light chain multiple myeloma with no measurable lesions in serum or urine: Serum free light chain ≥10 mg/dL and abnormal serum free light chain κ/γ ratio.

  6. The patient has recovered from toxicities associated with previous treatment, i.e., CTCAE toxicity grade <2 (unless the abnormality is related to the tumor or stable, with no significant impact on safety or efficacy as determined by the investigator).

  7. ECOG performance status of 0-2 and an expected survival of more than 3 months.

  8. Adequate organ function:
* Alanine transaminase (ALT) ≤3 times the upper limit of normal (ULN);
* Aspartate transaminase (AST) ≤3 times ULN;
* Total bilirubin ≤1.5 times ULN;
* Serum creatinine ≤1.5 times ULN, or creatinine clearance ≥60 mL/min;
* Indoor oxygen saturation ≥92%;
* Left ventricular ejection fraction (LVEF) ≥45%, confirmed by echocardiography with no clinically significant pericardial effusion or clinically significant electrocardiogram findings;
* No clinically significant pleural effusion. 9. Able to establish the required venous access for sample collection, with no contraindications for white blood cell collection.

Exclusion Criteria:

* 1. Diagnosed with or treated for invasive malignant tumors other than multiple myeloma.

  2. Previously received anti-tumor treatments including targeted therapy, epigenetic therapy, experimental drug therapy, or invasive experimental medical devices within 14 days or at least 5 half-lives (whichever is shorter) before the collection and preparation of CAR-T cells. Also, received monoclonal antibody therapy for relapsed/refractory multiple myeloma within 21 days, received cytotoxic therapy within 14 days, received proteasome inhibitor therapy within 14 days, received immunomodulatory agent therapy within 7 days, or received radiation therapy within 14 days (except for bone marrow reserves with field coverage ≤5%).

  3. Suspected involvement of multiple myeloma in the central nervous system or meninges confirmed by MRI or CT, or presence of other active central nervous system diseases.

  4. Screening criteria include plasma cell leukemia (according to standard classification, plasma cells >2.0×109/L), Waldenstrom macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or secondary AL amyloidosis.

  5. Positive for hepatitis B surface antigen (HBsAg) and positive for HBV-DNA; positive for hepatitis C virus (HCV) antibody; positive for human immunodeficiency virus (HIV) antibody; cytomegalovirus (CMV) DNA test result ≥500 copies/mL; positive for syphilis test.

  6. Positive for hepatitis C virus (HCV) antibody; positive for human immunodeficiency virus (HIV) antibody; cytomegalovirus (CMV) DNA test result ≥500 copies/mL; positive for syphilis test.

  7. History of severe allergies defined as grade II or above reactions, with clinical manifestations including airway obstruction (runny nose, coughing, wheezing, difficulty breathing), tachycardia, hypotension, arrhythmia, gastrointestinal symptoms (nausea, vomiting), urinary or fecal incontinence, laryngeal edema, bronchospasm, cyanosis, shock, respiratory or cardiac arrest, or known allergy to any active ingredient, excipient, murine-derived product, or xenogeneic protein contained in this trial (including the CleenRx regimen).

  8. Severe cardiac diseases including but not limited to severe arrhythmias, unstable angina pectoris, extensive myocardial infarction, New York Heart Association Class III or IV heart failure, myocardial infarction within 6 months before screening or coronary artery bypass graft (CABG), unexplained history of syncope unrelated to vasovagal or dehydration, severe non-ischemic cardiomyopathy, or uncontrolled hypertension (defined as failure to achieve blood pressure goals despite using ≥3 antihypertensive drugs, including diuretics, for ≥1 month or effective blood pressure control requiring ≥4 antihypertensive drugs).

  9. Unstable systemic diseases, including but not limited to severe liver, kidney, or metabolic diseases requiring medication.

  10. Acute/chronic graft-versus-host disease (GVHD) within 6 months before screening or patients requiring immunosuppressive therapy for GVHD.

  11. Active autoimmune or inflammatory diseases of the nervous system (e.g., Guillain-Barré syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular diseases (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES)).

  12. Presence of tumor emergencies (e.g., spinal cord compression, intestinal obstruction, leukostasis, tumor lysis syndrome) requiring urgent treatment during screening or before cell infusion.

  13. Uncontrolled bacterial, fungal, viral, or other infections requiring antibiotic treatment.

  14. Underwent major surgery (excluding diagnostic surgery and biopsies) within 4 weeks before CleenRx or planned major surgery during the study, or incomplete healing of surgical wounds before enrollment.

  15. Received (attenuated) live virus vaccines within 4 weeks before screening. 16. Presence of severe mental disorders. 17. Alcohol or substance abuse history. 18. Pregnant or breastfeeding women, and female subjects or male subjects with partners planning pregnancy within 2 years after cell infusion, and subjects who plan to become pregnant within 2 years after cell infusion. Additionally, according to the investigator's judgment and/or clinical criteria, patients with contraindications to any study procedures or other medical conditions that may expose them to unacceptable risks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-29 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Day 0, Month 1.5, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 18, Month 24
  Subjects were evaluated for efficacy according to the IMWG Efficacy Assessment Criteria (2016 revision).

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhang, Doctoral, Principal Investigator — Guangdong Second Provincial General Hospital
Locations (1):
- Guangdong Second Provincial General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chen D, You F, Xiang S, Wang Y, Li Y, Meng H, An G, Zhang T, Li Z, Jiang L, Wu H, Sheng B, Zhang B, Yang L. Chimeric antigen receptor T cells derived from CD7 nanobody exhibit robust antitumor potential against CD7-positive malignancies. Am J Cancer Res. 2021 Nov 15;11(11):5263-5281. eCollection 2021. PMID 34873460
- [Background] Benmebarek MR, Karches CH, Cadilha BL, Lesch S, Endres S, Kobold S. Killing Mechanisms of Chimeric Antigen Receptor (CAR) T Cells. Int J Mol Sci. 2019 Mar 14;20(6):1283. doi: 10.3390/ijms20061283. PMID 30875739
- [Background] Harris DT, Kranz DM. Adoptive T Cell Therapies: A Comparison of T Cell Receptors and Chimeric Antigen Receptors. Trends Pharmacol Sci. 2016 Mar;37(3):220-230. doi: 10.1016/j.tips.2015.11.004. Epub 2015 Dec 17. PMID 26705086
- [Background] Srivastava S, Riddell SR. Engineering CAR-T cells: Design concepts. Trends Immunol. 2015 Aug;36(8):494-502. doi: 10.1016/j.it.2015.06.004. Epub 2015 Jul 11. PMID 26169254
- [Background] Dotti G, Gottschalk S, Savoldo B, Brenner MK. Design and development of therapies using chimeric antigen receptor-expressing T cells. Immunol Rev. 2014 Jan;257(1):107-26. doi: 10.1111/imr.12131. PMID 24329793
- [Background] Neelapu SS, Locke FL, Bartlett NL, Lekakis LJ, Miklos DB, Jacobson CA, Braunschweig I, Oluwole OO, Siddiqi T, Lin Y, Timmerman JM, Stiff PJ, Friedberg JW, Flinn IW, Goy A, Hill BT, Smith MR, Deol A, Farooq U, McSweeney P, Munoz J, Avivi I, Castro JE, Westin JR, Chavez JC, Ghobadi A, Komanduri KV, Levy R, Jacobsen ED, Witzig TE, Reagan P, Bot A, Rossi J, Navale L, Jiang Y, Aycock J, Elias M, Chang D, Wiezorek J, Go WY. Axicabtagene Ciloleucel CAR T-Cell Therapy in Refractory Large B-Cell Lymphoma. N Engl J Med. 2017 Dec 28;377(26):2531-2544. doi: 10.1056/NEJMoa1707447. Epub 2017 Dec 10. PMID 29226797
- [Background] Schuster SJ, Bishop MR, Tam CS, Waller EK, Borchmann P, McGuirk JP, Jager U, Jaglowski S, Andreadis C, Westin JR, Fleury I, Bachanova V, Foley SR, Ho PJ, Mielke S, Magenau JM, Holte H, Pantano S, Pacaud LB, Awasthi R, Chu J, Anak O, Salles G, Maziarz RT; JULIET Investigators. Tisagenlecleucel in Adult Relapsed or Refractory Diffuse Large B-Cell Lymphoma. N Engl J Med. 2019 Jan 3;380(1):45-56. doi: 10.1056/NEJMoa1804980. Epub 2018 Dec 1. PMID 30501490
- [Background] Maude SL, Laetsch TW, Buechner J, Rives S, Boyer M, Bittencourt H, Bader P, Verneris MR, Stefanski HE, Myers GD, Qayed M, De Moerloose B, Hiramatsu H, Schlis K, Davis KL, Martin PL, Nemecek ER, Yanik GA, Peters C, Baruchel A, Boissel N, Mechinaud F, Balduzzi A, Krueger J, June CH, Levine BL, Wood P, Taran T, Leung M, Mueller KT, Zhang Y, Sen K, Lebwohl D, Pulsipher MA, Grupp SA. Tisagenlecleucel in Children and Young Adults with B-Cell Lymphoblastic Leukemia. N Engl J Med. 2018 Feb 1;378(5):439-448. doi: 10.1056/NEJMoa1709866. PMID 29385370
- [Background] Rodriguez-Lobato LG, Ganzetti M, Fernandez de Larrea C, Hudecek M, Einsele H, Danhof S. CAR T-Cells in Multiple Myeloma: State of the Art and Future Directions. Front Oncol. 2020 Jul 28;10:1243. doi: 10.3389/fonc.2020.01243. eCollection 2020. PMID 32850376
- [Background] Munshi NC, Anderson LD Jr, Shah N, Madduri D, Berdeja J, Lonial S, Raje N, Lin Y, Siegel D, Oriol A, Moreau P, Yakoub-Agha I, Delforge M, Cavo M, Einsele H, Goldschmidt H, Weisel K, Rambaldi A, Reece D, Petrocca F, Massaro M, Connarn JN, Kaiser S, Patel P, Huang L, Campbell TB, Hege K, San-Miguel J. Idecabtagene Vicleucel in Relapsed and Refractory Multiple Myeloma. N Engl J Med. 2021 Feb 25;384(8):705-716. doi: 10.1056/NEJMoa2024850. PMID 33626253
- [Background] Rabinowich H, Pricop L, Herberman RB, Whiteside TL. Expression and function of CD7 molecule on human natural killer cells. J Immunol. 1994 Jan 15;152(2):517-26. PMID 7506726